CLINICAL TRIAL: NCT05309681
Title: Salivary Melatonin Levels and Sleep Quality in Patients With Burning Mouth Syndrome
Status: Completed | Type: Observational
Sponsor: University of Zagreb (Other)
Responsible Party: Principal Investigator, Božana Lončar Brzak, Assistant Professor at the Department of Oral Medicine, University of Zagreb
Other Study IDs: 09/2020
Record Dates: First submitted 2022-03-24; First posted 2022-04-04 (Actual); Last update posted 2022-05-25 (Actual); Status verified 2022-05

CONDITIONS: Burning Mouth Syndrome; Melatonin
MeSH Terms: conditions — Burning Mouth Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — unstimulated saliva samples
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study group: Female patients of the Department of Oral medicine diagnosed with burning mouth syndrome
  Interventions: Other: Epworth's sleepiness scale; unstimulated saliva sample
- Control group: Age-matched female patients without oral lesions and without burning mouth syndrome
  Interventions: Other: Epworth's sleepiness scale; unstimulated saliva sample

INTERVENTIONS:
Other: Epworth's sleepiness scale; unstimulated saliva sample — Unstimulated saliva sample; Epworth's sleepiness scale

SUMMARY:
Burning mouth syndrome is an idiopathic condition characterized by symptoms burning and / or pain of the oral mucosa with an orderly clinical finding. So far not found a unique way of treatment. It is a diagnosis that impairs the quality of life of patients, and consequently it can affect the quality of sleep. Melatonin is a hormone secreted from pineal gland and regulates the day-night rhythm of man, and whose production in the body decreases aging. The level of melatonin in saliva correlates well with the level of melatonin in plasma, therefore they are advantages of determining from saliva painlessness and non-invasiveness of the procedure itself. The purpose of this study was to compare the level of melatonin in saliva and the quality of sleep with help of the Epworth Sleepiness Scale in patients with burning mouth syndrome and control groups of patients without subjective oral disorders and with an orderly clinical finding.

ELIGIBILITY:
Inclusion Criteria:

* female patients
* primary burning mouth syndrome
* without oral lesions

Exclusion Criteria:

* secondary burning mouth syndrome
* male gender
* patients with oral lesions

Ages: 18 Years to 65 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Female patients with burning mouth syndrome and age-matched female controls without burning mouth syndrome or oral lesions will be included in the study. A sample of unstimulated saliva will be taken from all patients and frozen. All patients will also fill in Epworth's sleepiness scale.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2021-01-07 (Actual); Primary Completion 2021-07-18 (Actual); Study Completion 2021-12-15 (Actual)

PRIMARY OUTCOMES:
determining the level of salivary melatonin | January 2021-July 2021
  The level of salivary melatonin will be determined in frozen samples of unstimulated saliva samples

SECONDARY OUTCOMES:
determining the difference in Epworth's sleepiness scale | January 2021-July 2021
  The test is a list of eight situations in which you rate your tendency to become sleepy on a scale of 0, no chance of dozing, to 3, high chance of dozing. Total score is graded from 0-24. 0-7:It is unlikely that you are abnormally sleepy.
  8-9:You have an average amount of daytime sleepiness. 10-15:You may be excessively sleepy depending on the situation. You may want to consider seeking medical attention. 16-24:You are excessively sleepy and should consider seeking medical attention.

CONTACTS AND LOCATIONS:
Locations (1):
- School of Dental Medicine, University of Zagreb, Zagreb, Croatia

IPD SHARING:
Plan to Share IPD: No